CLINICAL TRIAL: NCT01706900
Title: Incubator Temperature for Culturing Human Embryos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Laboratory Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IbnSina Hospital
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Embryo Culture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incubator Temp 37 degree (Placebo Comparator): We will set incubator Temp to 37 degree as the routine embryo culture Temp since 1978 as the placebo arm.
  Interventions: Other: Incubator Temp 37 degree
- Incubator Temp set to 36.5 degree (Experimental): We will set incubator Temp to 36.5 so we can assess the outcome and compare the results with the placebo group.
  Interventions: Other: Incubator Temp set to 36.5 degree

INTERVENTIONS:
Other: Incubator Temp set to 36.5 degree — We will set incubator Temp to 36.5 so we can assess the outcome and compare the results with the placebo group.
  Arms: Incubator Temp set to 36.5 degree
Other: Incubator Temp 37 degree — We will set incubator Temp to 37 degree as the routine embryo culture Temp since 1978 as the placebo arm.
  Arms: Incubator Temp 37 degree

SUMMARY:
Incubator temperature is one of the most precious variables in IVF labs. When the IVF started, almost all incubator temperatures were set at 37 degrees which mimic in vivo conditions. Some authors speculated that gametes and early embryos might need low temperatures that provide quieter metabolism. We decide to compare Embryo culture at 37 degree or slightly lower 36.5 degree and extensively investigate to find which is better to crucially introduce a solid evidence through this RCT.

DETAILED DESCRIPTION:
Since the first IVF birth in 1978, the field of assisted reproductive technology has evolved dramatically. The evolution includes both the ovarian stimulation protocols and the laboratory techniques. Optimization of the laboratory procedures is of great interest to the scientists in the field of IVF.

Incubator temperature is one of the most precious variables in IVF labs. When the IVF started, almost all incubator temperatures were set at 37 degrees which mimic in vivo conditions.

Some authors speculated that gametes and early embryos might need low temperatures that provide quieter metabolism. another group found increase in pregnancy rate for embryos cultured below 37 degree compared to those cultured at 37 degree. Nevertheless; the majority of embryologists still consider culture at 37 degrees is the back bone for the incubators.

The paucity of well designed studies makes it difficult to achieve a satisfactory answer whether lower temperature will improve the pregnancy rate. This encourage us to study the effect of lower temperature (36.5 degrees) on the pregnancy rate compared to conventional temperature (37 degrees).

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≤ 33 years
* BMI ≤ 33
* Normal responder ( ≥ 8 MII )
* Fresh cycle
* First attempt (or with previous successful attempt)
* Normal or mild oligoasthenoteratozoospermia

Exclusion Criteria:

* Testicular sperm
* < 8 MIII collected
* Difficult transfer cycle
* endometriotic patients
* Poor Endometrium < 8mm diameter at OPU

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fetal heart beat rate | 3 months
  Compare the fetal heart beat rate between the 2 study arms in the first 3 months following Embryo Transfer.

SECONDARY OUTCOMES:
Pregnancy rate | one month
  Measure the pregnancy rate between the 2 study arms in the following one month after Embryo Transfer
Top quality embryos Day3 | one week
  Measure the top quality embryos day3 between the 2 study arms in the following week after ICSI
blastocyst formation rate | one week
  Measure the blastocyst formation rate between the 2 study arms in the following week after ICSI
Top quality blastocyst | one week
  Measure the top quality blastocyst rate between the 2 study arms in the following week after ICSI
Implantation rate | one month
  Measure the implantation rate between the 2 study arms in the following first month after Embryo Transfer

OTHER OUTCOMES:
Cleavage rate on day 3 | one month
  We will measure the rate of embryo cleavage on day3 between the 2 study arms

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad F. Abdel-Raheem, Lab Director, Principal Investigator — IbnSina IVF Center; Mohamed Y. Abdel-Rahman, M.D., Principal Investigator — IbnSina IVF center; Hesham A. Kasem, Gynaecologist, Principal Investigator — IbnSina IVF Center
Locations (1):
- IbnSina IVF Center, IbnSina Hospital, Sohag, Sohag Governorate, Egypt